CLINICAL TRIAL: NCT02988869
Title: Comparison of Bronchodilator Efficacy of Tiotropium/Formoterol Combination Treatment Administered (qd) Via Discair® With Tiotropium (qd) Monotherapy or Tiotropium (qd) + Formoterol (Bid) Free Combination Treatment in Patients With Chronic Obstructive Pulmonary Disease (COPD)
Brief Title: Tiotropium/Formoterol Via Discair® vs Tiotropium Monotherapy or Tiotropium + Formoterol Free Combination Treatment
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Neutec Ar-Ge San ve Tic A.Ş (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NEU-22.12
Record Dates: First submitted 2016-10-06; First posted 2016-12-09 (Estimated); Last update posted 2020-06-16 (Actual); Status verified 2017-12

CONDITIONS: COPD
Keywords: COPD; Tiotropium; Formoterol
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Tiotropium Bromide; Formoterol Fumarate; Neptune

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Tiotropium/Formoterol (Experimental): Tiotropium/Formoterol 18/12 mcg Inhalation Powder (1 puff) once daily via Discair®
  Interventions: Drug: Tiotropium/Formoterol
- Tiotropium (Active Comparator): Tiotropium 18 mcg Inhalation Powder (1 puff) once daily via Handihaler
  Interventions: Drug: Tiotropium
- Tiotropium + Formoterol (Active Comparator): Tiotropium 18 mcg Inhalation Powder (1 puff) once daily via Handihaler + Formoterol 12 mcg Inhalation Powder (1 puff) twice daily via Aerolizer
  Interventions: Drug: Formoterol; Drug: Tiotropium

INTERVENTIONS:
Drug: Tiotropium/Formoterol — Tiotropium/Formoterol 18/12 mcg Inhalation Powder (1 puff) once daily via Discair®
  Other Names: TRITON 18/12 mcg Discair Inhalation Powder
  Arms: Tiotropium/Formoterol
Drug: Tiotropium — Tiotropium 18 mcg Inhalation Powder (1 puff) once daily via Handihaler
  Other Names: SPIRIVA 18 mcg Inhalation Powder
  Arms: Tiotropium
Drug: Formoterol — Formoterol 12 mcg Inhalation Powder (1 puff) twice daily via Aerolizer
  Other Names: FORADIL 12 mcg Inhalation Powder
  Arms: Tiotropium + Formoterol
Drug: Tiotropium — Tiotropium 18 mcg Inhalation Powder (1 puff) once daily via Handihaler
  Other Names: SPIRIVA Inhalation Powder
  Arms: Tiotropium + Formoterol

SUMMARY:
The overall objective is to asses the bronchodilator effect of once daily Tiotropium/Formoterol combination delivered via Discair® by comparing Tiotropium (q.d.) monotherapy delivered via Handihaler and tiotropium (q.d.) delivered via Handihaler + formoterol (b.i.d) delivered via Aerolizer free combination treatment in patients with stable moderate to severe COPD.

Spirometric measurements (FEV1, FVC) will be performed for a period of 24 h at 12 different times: pre-treatment (15 min prior to the first dose) and post-treatment (30. min, 60 min [1 hr], 120 min [2 hr], 180 min [3 hr], 240 min [4 hr], 360 min [6 hr], 480 min [8 hr], 600 min [10 hr], 720 min [12 hr], 840 min [14 hr],1440 min [24 hr].

DETAILED DESCRIPTION:
The overall objective is to asses the bronchodilator effect of once daily Tiotropium/Formoterol combination delivered via Discair® by comparing Tiotropium (q.d.) monotherapy delivered via Handihaler and tiotropium (q.d.) delivered via Handihaler + formoterol (b.i.d) delivered via Aerolizer free combination treatment in patients with stable moderate to severe COPD.

Patients will be randomly assigned to receive Tiotropium/Formoterol combination as dry powder for inhalation by Discair® (test inhaler, n = 29) or Tiotropium as dry powder capsule for inhalation by HandiHaler or tiotropium dry powder capsule for inhalation by HandiHaler + formoterol as dry powder capsule for inhalation by Aerolizer. Patients will be evaluated at 4 consecutive visits: baseline (enrollment), screening, treatment, and 24h after treatment.

For newly diagnosed and formerly diagnosed patients who are not on COPD medication, the screening visit will be performed on the day of enrollment. For formerly diagnosed patients receiving COPD treatment, the day of the screening visit will be based on the completion of a run-in period, with the length determined by the specific medication. During the run-in period, salbutamol (100 µg inhaler) will be prescribed as a rescue medication.

Spirometric measurements (FEV1, FVC) will be performed for a period of 24 h at 12 different times: pre-treatment (15 min prior to the first dose) and post-treatment (30. min, 60 min [1 hr], 120 min [2 hr], 180 min [3 hr], 240 min [4 hr], 360 min [6 hr], 480 min [8 hr], 600 min [10 hr], 720 min [12 hr], 840 min [14 hr],1440 min [24 hr].

ELIGIBILITY:
Inclusion Criteria:

* Patients aged ≥40 years with COPD diagnosis according to the current GOLD (The Global Initiative for Chronic Obstructive Lung Disease) strategy.
* Patients who have symptomatic stable moderate to severe COPD diagnosis with post-bronchodilator FEV1/FVC ratio <0.70, and FEV1 <80% of predicted normal at screening visit.
* Current smokers or ex-smokers with a smoking history of at least 10 pack-years
* Patients who have no exacerbation within last 4 weeks
* Female patients with childbearing potential using effective birth control method
* Patients who signed written informed consent prior to participation
* Patients who accept to comply with the requirements of the protocol
* Patients who have a capability of communicate with investigator

Exclusion Criteria:

* History of hypersensitivity to drugs contains anticholinergics, beta-adrenergic, lactose
* Diagnosis of asthma
* Patients vaccinated with live attenuated vaccines within 2 weeks prior to screening visit or during run-in period.
* Patients who had COPD exacerbation or lower respiratory track infections that required antibiotic, oral or parenteral corticosteroid treatment within 4 weeks prior to screening visit or during run-in period.
* Patients who have a history of myocardial infarction, hearth failure, acute ischemic coroner disease or severe cardiac arrhythmia requiring treatment within least 6 weeks
* Patients who have lung cancer
* Patients with active tuberculosis
* Patients who use oxygen therapy
* Patients who have common interstitial lung diseases like cystic fibrosis, bronchiolitis obliterans
* Patients with serious liver or renal disease that leads to organ failure
* Women who are pregnant or nursing
* History of allergic rhinitis and atopy
* Known symptomatic prostatic hypertrophy requiring drug therapy or operation
* Patients with narrow-angle glaucoma requiring drug therapy

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Actual)
Dates: Start 2016-08 (Actual); Primary Completion 2017-08 (Actual); Study Completion 2017-08 (Actual)

PRIMARY OUTCOMES:
Mean max change (ml) from baseline in FEV1 over a period of 24 h. | Pre-treatment (10 minutes prior to the first dose of randomized study medication) and post-treatment (Day 1)
  Spirometric measurements will be made at 10 minutes prior to the first dose of randomized study medication and and post-treatment at 30. min, 60 min, 120 min, 180 min, 240 min, 360 min, 480 min, 600 min, 720 min, 840 min, 1440 min.
Mean % change from baseline in FEV1 over a period of 24 h. | Pre-treatment (10 minutes prior to the first dose of randomized study medication) and post-treatment (Day 1)
  Spirometric measurements will be made at 10 minutes prior to the first dose of randomized study medication and and post-treatment at 30. min, 60 min, 120 min, 180 min, 240 min, 360 min, 480 min, 600 min, 720 min, 840 min, 1440 min.
Mean max change (ml) from baseline in FVC over a period of 24 h. | Pre-treatment (10 minutes prior to the first dose of randomized study medication) and post-treatment (Day 1)
  Spirometric measurements will be made at 10 minutes prior to the first dose of randomized study medication and and post-treatment at 30. min, 60 min, 120 min, 180 min, 240 min, 360 min, 480 min, 600 min, 720 min, 840 min, 1440 min.
Mean % change from baseline in FVC over a period of 24 h. | Pre-treatment (10 minutes prior to the first dose of randomized study medication) and post-treatment (Day 1)
  Spirometric measurements will be made at 10 minutes prior to the first dose of randomized study medication and and post-treatment at 30. min, 60 min, 120 min, 180 min, 240 min, 360 min, 480 min, 600 min, 720 min, 840 min, 1440 min.
FEV1 (AUC0-12) response | From pre-treatment (10 minutes prior to the first dose of randomized study medication) to 12 hours post-treatment (Day 1)
  Spirometric measurements will be made at 10 minutes prior to the first dose of randomized study medication and and post-treatment at 30. min, 60 min, 120 min, 180 min, 240 min, 360 min, 480 min, 600 min, 720 min, 840 min, 1440 min.
FVC (AUC0-12) response | From pre-treatment (10 minutes prior to the first dose of randomized study medication) to 12 hours post-treatment (Day 1)
  Spirometric measurements will be made at 10 minutes prior to the first dose of randomized study medication and and post-treatment at 30. min, 60 min, 120 min, 180 min, 240 min, 360 min, 480 min, 600 min, 720 min, 840 min, 1440 min.
FEV1 (AUC0-24) response | From pre-treatment (10 minutes prior to the first dose of randomized study medication) to 24 hours post-treatment (Day 1)
  Spirometric measurements will be made at 10 minutes prior to the first dose of randomized study medication and and post-treatment at 30. min, 60 min, 120 min, 180 min, 240 min, 360 min, 480 min, 600 min, 720 min, 840 min, 1440 min.
FVC (AUC0-24) response | From pre-treatment (10 minutes prior to the first dose of randomized study medication) to 24 hours post-treatment (Day 1)
  Spirometric measurements will be made at 10 minutes prior to the first dose of randomized study medication and and post-treatment at 30. min, 60 min, 120 min, 180 min, 240 min, 360 min, 480 min, 600 min, 720 min, 840 min, 1440 min.
FEV1 (AUC12-24) response | From pre-treatment (10 minutes prior to the first dose of randomized study medication) to 24 hours post-treatment (Day 1)
  Spirometric measurements will be made at 10 minutes prior to the first dose of randomized study medication and and post-treatment at 30. min, 60 min, 120 min, 180 min, 240 min, 360 min, 480 min, 600 min, 720 min, 840 min, 1440 min.
FVC (AUC12-24) response | From pre-treatment (10 minutes prior to the first dose of randomized study medication) to 24 hours post-treatment (Day 1)
  Spirometric measurements will be made at 10 minutes prior to the first dose of randomized study medication and and post-treatment at 30. min, 60 min, 120 min, 180 min, 240 min, 360 min, 480 min, 600 min, 720 min, 840 min, 1440 min.

SECONDARY OUTCOMES:
The time to onset of bronchodilator effect | Pre-treatment (10 minutes prior to the first dose of randomized study medication) and post-treatment (Day 1)
  Spirometric measurements will be made at 10 minutes prior to the first dose of randomized study medication and and post-treatment at 30. min, 60 min, 120 min, 180 min, 240 min, 360 min, 480 min, 600 min, 720 min, 840 min, 1440 min.
The time to onset of maximum effect | Pre-treatment (10 minutes prior to the first dose of randomized study medication) and post-treatment (Day 1)
  Spirometric measurements will be made at 10 minutes prior to the first dose of randomized study medication and and post-treatment at 30. min, 60 min, 120 min, 180 min, 240 min, 360 min, 480 min, 600 min, 720 min, 840 min, 1440 min.
Evaluation of safety (Physical examination, numbers of adverse reactions and abnormal laboratory values related to treatment) | Predose and up to 24 hours postdose

CONTACTS AND LOCATIONS:
Overall Officials: Pinar Yildiz, Professor Doctor, Principal Investigator — Yedikule Chest Diseases and Thoracic Surgery Training and Research Hospital-Turkey
Locations (1):
- Yedikule Chest Diseases and Thoracic Surgery Training and Research Hospital, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Yildiz BP, Bayraktaroglu M, Gunen H. Bronchodilator efficacy of tiotropium/formoterol (18/12 microg once daily via a Discair inhaler), tiotropium alone (18 microg by Handihaler) or combined with formoterol (12 microg twice daily by Aerolizer) in adults with moderate-to-severe stable COPD. Curr Med Res Opin. 2019 Dec;35(12):2187-2196. doi: 10.1080/03007995.2019.1654722. Epub 2019 Sep 16. PMID 31397184
- [Result] Yildiz BP, Bayraktaroglu M, Gunen H. Reply: Re: Yildiz BP, Bayraktaroglu M, Gunen H. Bronchodilator efficacy of tiotropium/formoterol (18/12 mug once daily via a discair inhaler), tiotropium alone (18 mug by handihaler) or combined with formoterol (12 mug twice daily by aerolizer) in adults with moderate-to-severe stable COPD. Curr Med Res Opin. 2019;35(12):2187-2196. Curr Med Res Opin. 2020 Jun;36(6):1061-1062. doi: 10.1080/03007995.2020.1754187. Epub 2020 Apr 29. No abstract available. PMID 32270722